CLINICAL TRIAL: NCT06138782
Title: Identifying Networks Underlying Compulsivity in Anorexia Nervosa for Targeting With Neuromodulation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-39333
Record Dates: First submitted 2023-10-09; First posted 2023-11-18 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Anorexia Nervosa
Keywords: anorexia; AN; anorexia nervosa; OCD; obsessive; obsessive-compulsive disorder
MeSH Terms: conditions — Anorexia Nervosa; Anorexia; Obsessive-Compulsive Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TMS (Aim 2) (Experimental): Our protocol consists of five treatments of inhibitory continuous TBS (cTBS) to the R OFC lasting three minutes delivered every hour over the course of 10 days (2 weeks) for a total of 50 treatments.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — Our protocol consists of five treatments of inhibitory continuous TBS (cTBS) to the R OFC lasting three minutes delivered every hour over the course of 10 days (2 weeks) for a total of 50 treatments.

SUMMARY:
Transcranial Magnetic Stimulation (TMS) is approved by the Food and Drug Administration (FDA) for the treatment of refractory Major Depressive Disorder (MDD) and obsessive-compulsive disorder (OCD). Anorexia nervosa (AN) is characterized by restrictive eating leading to low weight and associated complications. There is an emerging understanding that the symptoms of OCD and AN overlap as AN can be characterized by obsessive thought patterns around food and compulsive restricting and weight loss behaviors. Both conditions are characterized by a propensity toward cognitive inflexibility and the conditions may share neural substrates that maintain maladaptive habitual behaviors and cognitive rigidity. An evidence-based repetitive transcranial magnetic stimulation (rTMS) target for OCD is the orbitofrontal cortex (OFC). The investigators intend to determine if the OFC is also a potential rTMS target for AN and to determine if there is a characteristic pattern of functional network reorganization as characterized by functional magnetic resonance imaging (fMRI) in TMS responders.

DETAILED DESCRIPTION:
To determine if accelerated theta burst rTMS can treat symptoms of AN and normalize abnormal network connectivity, the investigators will enroll 20 patients with AN (aged 16-45) to receive five treatments of inhibitory continuous theta burst rTMS to the right orbitofrontal cortex (R OFC) lasting three minutes delivered every hour over the course of 10 days (2 weeks) for a total of 50 treatments, with follow-up immediately post-treatment, and at 1 month. Clinical symptom change will be determined with weight gain from percent expected body weight (%EBW) and clinical interview with the Eating Disorders Examination (EDE) as well as validated self-report. For Hypothesis 1: At 1-month post-rTMS, the investigators expect increased %EBW, and meaningful reductions in AN compulsive symptoms per the EDE. For Hypothesis 2: The investigators intend to identify changes in the default mode network comparing before and after TMS that are associated with an improvement in AN compulsive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* outpatients
* ages 16 - 75 for Aim 2
* meets Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for AN
* stable on chronic psychotropic medications for 4 weeks prior to the study and agreeable to continue throughout the study
* participants may continue to take medications and record daily usage throughout the study
* capacity to provide informed consent
* ability to tolerate clinical study procedures
* successfully complete the screening forms without any contraindications

Exclusion Criteria:

* Psychiatric: schizophrenia, bipolar disorder, prior psychosurgery, prior electroconvulsive therapy (ECT)
* Neurologic: severe neurocognitive disorder, seizure disorder, certain structural brain lesions (e.g., intracranial mass lesions, hydrocephalus, sequelae of meningitis)
* TMS contraindications: implanted device; presence of metal in the head, including eyes and ears (excluding dental implants); certain tics; medications or systemic illness that predispose seizure risk
* Subjects with an unstable physical, systemic, or metabolic disorder (e.g., unstable hypertension)
* Females who are pregnant or nursing
* Inability to complete the research study

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Eating Disorders Examination - Questionnaire (EDE-Q) | Baseline; day 1, 5, & 10 of TMS; every follow-up (weeks 1, 2, & 3 after final TMS treatment; every month for a year).
  The Eating Disorder Examination Questionnaire (EDE-Q) is a 28-item self-report questionnaire designed to assess the range, frequency and severity of behaviours associated with a diagnosis of an eating disorder. It is categorised into 4 subscales (Restraint, Eating Concern, Shape Concern and Weight Concern) and an overall global score, with a higher score indicating more problematic eating difficulties.

SECONDARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale (Y-BOCS) | Baseline; all 10 days of TMS; every follow-up (weeks 1, 2, & 3 after final TMS treatment; every month for a year).
  The Y-BOCS is a 10-item ordinal scale (0-4) that rates the severity separately for both obsessions and compulsions of OCD according to the time occupied, degree of interference, subjective distress, internal resistance, and degree of control. Higher scores indicate worse outcome.
Compulsive Exercise Test (CET) | Baseline; day 1, 5, & 10 of TMS; every follow-up (weeks 1, 2, & 3 after final TMS treatment; every month for a year).
  The CET is a 24-item self-report measure designed to assess the core features of excessive exercise in the eating disorders. Higher scores indicate worse outcome.
State Trait Anxiety Index (STAI) | Baseline; all 10 days of TMS; every follow-up (weeks 1, 2, & 3 after final TMS treatment; every month for a year).
  The Spielberger State-Trait Anxiety Inventory (STAI) is a 40-item self-report measure of anxiety using a 4-point Likert-type scale (from 0 to 3 points) for each item. It has two scales: State anxiety, i.e. how one feels at the moment; and Trait anxiety, i.e. how one generally feels. Higher scores indicate worse outcome.
Ecological Momentary Assessment (EMA) | Baseline; all 10 days of TMS; every follow-up (weeks 1, 2, & 3 after final TMS treatment; every month for a year).
  Ecological momentary assessments (EMAs) study people's thoughts and behavior in their daily lives by repeatedly collecting data in an individual's normal environment, at or close to the time that the individual carries out that behavior. Higher scores indicate worse outcome.
Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline; all 10 days of TMS; every follow-up (weeks 1, 2, & 3 after final TMS treatment; every month for a year).
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Higher scores indicate worse outcome.
Hamilton Self-Rating Scale for Depression (HAM-D) | Baseline; all 10 days of TMS; every follow-up (weeks 1, 2, & 3 after final TMS treatment; every month for a year).
  The HAM-D is a multiple-item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery. Higher scores indicate worse outcome.
Intolerance of Uncertainty Scale - short form (IUS-12) | Baseline; all 10 days of TMS; every follow-up (weeks 1, 2, & 3 after final TMS treatment; every month for a year).
  The Intolerance of Uncertainty Scale (IUS) includes items relating to the idea that uncertainty is unacceptable, reflects badly on a person, and leads to frustration, stress, and the inability to take action. Higher scores indicate worse outcome.
Repetitive Thinking Questionnaire-10 (RTQ-10) | Baseline; all 10 days of TMS; every follow-up (weeks 1, 2, & 3 after final TMS treatment; every month for a year).
  The Repetitive Thinking Questionnaire (RTQ) was developed by combining items from commonly used measures of worry, rumination, and post-event processing, and then modifying the items to remove diagnosis-specific content. It is used to measure repetitive negative thinking. Higher scores indicate worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Lee, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carmi L, Tendler A, Bystritsky A, Hollander E, Blumberger DM, Daskalakis J, Ward H, Lapidus K, Goodman W, Casuto L, Feifel D, Barnea-Ygael N, Roth Y, Zangen A, Zohar J. Efficacy and Safety of Deep Transcranial Magnetic Stimulation for Obsessive-Compulsive Disorder: A Prospective Multicenter Randomized Double-Blind Placebo-Controlled Trial. Am J Psychiatry. 2019 Nov 1;176(11):931-938. doi: 10.1176/appi.ajp.2019.18101180. Epub 2019 May 21. PMID 31109199
- [Background] Graybiel AM, Rauch SL. Toward a neurobiology of obsessive-compulsive disorder. Neuron. 2000 Nov;28(2):343-7. doi: 10.1016/s0896-6273(00)00113-6. No abstract available. PMID 11144344
- [Background] Kaye W. Is food restriction in anorexia nervosa caused by reduced reward and/or increased inhibition? Neuropsychopharmacology. 2011;36(Kaye W.) UCSD, Department of Psychiatry, San Diego, United States):S48. doi:10.1038/npp.2011.290
- [Background] Kaye WH, Bulik CM. Treatment of Patients With Anorexia Nervosa in the US-A Crisis in Care. JAMA Psychiatry. 2021 Jun 1;78(6):591-592. doi: 10.1001/jamapsychiatry.2020.4796. No abstract available. PMID 33625500
- [Background] Murray SB, Strober M, Craske MG, Griffiths S, Levinson CA, Strigo IA. Fear as a translational mechanism in the psychopathology of anorexia nervosa. Neurosci Biobehav Rev. 2018 Dec;95:383-395. doi: 10.1016/j.neubiorev.2018.10.013. Epub 2018 Oct 28. PMID 30392878
- [Background] Nauczyciel C, Le Jeune F, Naudet F, Douabin S, Esquevin A, Verin M, Dondaine T, Robert G, Drapier D, Millet B. Repetitive transcranial magnetic stimulation over the orbitofrontal cortex for obsessive-compulsive disorder: a double-blind, crossover study. Transl Psychiatry. 2014 Sep 9;4(9):e436. doi: 10.1038/tp.2014.62. PMID 25203167
- [Background] Posner J, Song I, Lee S, Rodriguez CI, Moore H, Marsh R, Blair Simpson H. Increased functional connectivity between the default mode and salience networks in unmedicated adults with obsessive-compulsive disorder. Hum Brain Mapp. 2017 Feb;38(2):678-687. doi: 10.1002/hbm.23408. Epub 2016 Sep 23. PMID 27659299
- [Background] Steward T, Menchon JM, Jimenez-Murcia S, Soriano-Mas C, Fernandez-Aranda F. Neural Network Alterations Across Eating Disorders: A Narrative Review of fMRI Studies. Curr Neuropharmacol. 2018;16(8):1150-1163. doi: 10.2174/1570159X15666171017111532. PMID 29046154
- [Background] Walsh BT, Xu T, Wang Y, Attia E, Kaplan AS. Time Course of Relapse Following Acute Treatment for Anorexia Nervosa. Am J Psychiatry. 2021 Sep 1;178(9):848-853. doi: 10.1176/appi.ajp.2021.21010026. Epub 2021 Jun 22. PMID 34154394
- [Background] Whitfield-Gabrieli S, Ford JM. Default mode network activity and connectivity in psychopathology. Annu Rev Clin Psychol. 2012;8:49-76. doi: 10.1146/annurev-clinpsy-032511-143049. Epub 2012 Jan 6. PMID 22224834